CLINICAL TRIAL: NCT02257983
Title: A Phase 2A Randomized, Placebo Controlled, Double Blind Study of the Protective Effects of EPI-743 (VincerinoneTM) on Noise-Induced Hearing Loss
Brief Title: Protective Effects of EPI-743 on Noise-Induced Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EPI743-14-026
Record Dates: First submitted 2014-08-11; First posted 2014-10-07 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Noise-induced Hearing Loss
Keywords: hearing; noise; oxidative stress
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EPI-743 (Active Comparator): EPI-743 400 mg P.O. TID
  Interventions: Drug: EPI-743
- Placebo (Placebo Comparator): Sesame Oil, NF in sealed gelatin capsules to match the test product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EPI-743 — EPI-743 (2 capsules 200 mg each) taken at a dose of 400 mg P.O. TID for 9 days with noise exposure for 4 hours on Day 8.
  Other Names: VincerinoneTM; EPI743
  Arms: EPI-743
Drug: Placebo — 2 Placebo capsules P.O. TID for 9 days with noise exposure for 4 hours on Day 8.
  Other Names: Matching placebo
  Arms: Placebo

SUMMARY:
If effective, administration of EPI-743 should have protective effects against temporary noise-induced hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults ages 18-30
* Abstention from use of Idebenone, CoQ10, Vitamin E and foods or beverages at least 30 days prior to treatment initiation
* Non-smokers
* Abstention from alcohol from day 0 and throughout the duration of study
* Normal audiology exam
* Subject must be able to swallow size 0 capsules

Exclusion Criteria:

* Allergy to EPI-743 or sesame oil or nuts
* Any medical disordere that would prevent subject participation
* Any prescription meds other than for contraception or seasonal allergies
* Any significant patient medical history (cancer, cardiovascular, pulmonary, cognitive, ADHD, hx. of migraines, neurological, kidney)
* Fat malabsorption syndromes
* Anticoagulation thereapy within 30 days of enrollment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Pure tone audiometry | 9 days

SECONDARY OUTCOMES:
Time to recovery following acute noise exposure | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Le Prell, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- See also: Related Info — http://www.edisonpharma.com